CLINICAL TRIAL: NCT00760968
Title: A Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Evaluate the Safety and Efficacy of Oral TAK-783 in the Treatment of the Signs and Symptoms in Subjects With Rheumatoid Arthritis
Brief Title: Efficacy and Safety of TAK-783 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: VP Clinical Science, Takeda Global Research & Development Centre (Europe) Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-783-EC201; 2006-003054-26 (EudraCT Number); U1111-1114-0266 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Drug Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-783 100 mg QD + Methotrexate (Experimental)
  Interventions: Drug: TAK-783 and methotrexate
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: TAK-783 and methotrexate — TAK-783 100 mg, tablets, orally, once daily and methotrexate stable dose therapy for up to 12 weeks.
  Other Names: Rheumatrex®.
  Arms: TAK-783 100 mg QD + Methotrexate
Drug: Methotrexate — TAK-783 placebo-matching tablets, orally, once daily and methotrexate stable dose therapy for up to 12 weeks.
  Other Names: Rheumatrex®.
  Arms: Methotrexate

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-783, once daily (QD), taken in combination with methotrexate in subjects with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis affects approximately 1% of the adult population. It is a chronic, progressive disease characterized by synovial inflammation. The resulting inflammation leads to destruction of the synovium and surrounding joint tissues, which can result in cartilage destruction, bone erosion and resultant loss of joint function. It is an autoimmune disorder of unknown etiology and typically affects the joints of the hand, wrist, knee, and foot, usually in a bilateral pattern. Symptoms experienced early in the disease process include pain, swelling, and tenderness of affected joints. As the disease progresses, many patients experience joint stiffness, weakness, fatigue, anorexia, and weight loss, and ultimately tissue damage and joint destruction. The severity of symptoms varies widely, ranging from annoyance to debilitation. Rheumatoid arthritis is a disease that primarily afflicts adults, with women being affected more often than men. Because rheumatoid arthritis is both chronic and destructive, it requires early diagnosis and aggressive treatment to minimize the morbidity associated with its progression, which can lead to deterioration in physical function and psychological and social well-being. The objectives of rheumatoid arthritis therapy are to reduce inflammation and to decrease the progression of articular damage. Disease-modifying antirheumatic drugs are used to accomplish these objectives.

During the past several years, rheumatologists have become increasingly aggressive in initiating treatment with disease-modifying antirheumatic drugs early in the course of rheumatoid arthritis in an attempt to prevent joint destruction. The gold standard of therapy has been methotrexate, which has been shown to be efficacious and safe, and appears to remain effective, even after many years of treatment. However, not all patients respond to methotrexate, and even patients who do respond most frequently have only a partial response (reduced signs and symptoms, but still active disease). As a result, many patients are treated with 2 or more disease-modifying antirheumatic drugs at the same time.

More recently, biologics (biotechnology drugs) have been introduced in the armamentarium against rheumatoid arthritis, based on an improved understanding of the role of the proinflammatory mediators, TNF-alpha, interleukin-1, and interleukin-6 in rheumatoid arthritis. Etanercept (Enbrel®), a soluble TNF-alpha type II receptor-human immunoglobulin fusion protein administered subcutaneously twice a week, infliximab (Remicade®), a chimeric human mouse monoclonal antibody against TNF-alpha, administered intravenously every 4 to 8 weeks along with weekly methotrexate, and adalimumab (Humira®), a human-derived recombinant immunoglobulin monoclonal antibody, administered subcutaneously every other week, are currently available for treatment of rheumatoid arthritis. They have demonstrated rapid and substantial improvement in rheumatoid arthritis, presumably by preventing the actions of TNF-alpha in the joint, thereby reducing the inflammatory and destructive consequences of TNF-alpha. Etanercept and infliximab have been granted Food and Drug Administration (FDA) approved indications for reducing signs and symptoms, inhibiting the progression of structural damage and improving physical function of patients with moderately to severely active rheumatoid arthritis. Adalimumab has been granted FDA approved indications for reducing signs and symptoms and inhibiting the progression of structural damage, and Anakinra (Kineret®), an interleukin-1 receptor antagonist administered subcutaneously daily, received FDA approval for reducing signs and symptoms.

TAK-783 is being developed as an orally administered compound for the treatment of rheumatoid arthritis. Total participation time for this study is 16 to 40 weeks. All subjects will remain on a stable dose of methotrexate throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Had a diagnosis of rheumatoid arthritis using American College of Rheumatology criteria of at least 6 months duration and less than or equal to 3 years.
* A female subject of childbearing potential who is sexually active must agree to use adequate contraception, and must be neither pregnant nor lactating from Screening and throughout the duration of the study.
* Had a physical examination that, in the investigator's opinion, reveals no clinically significant abnormalities (other than rheumatoid arthritis), at the Screening Visit.
* Had clinical laboratory test results that are normal or, if abnormal, are not clinically significant in the investigator's opinion, at the Screening and Baseline Visits.
* Had a 12-lead electrocardiogram that is normal during the Screening Period, or, if abnormal, is not clinically significant in the opinion of the investigator.
* Had a chest x-ray within 3 months prior to or during the Pretreatment Period that, in the opinion of the investigator, is free of clinically significant findings.
* Had a negative purified protein derivative skin test for tuberculosis (less than or equal to 5 mm in duration) at screening and a negative tuberculosis screening history.
* Was receiving oral or parenteral methotrexate for at least 6 months prior to the Baseline Visit, and must be on a stable dose of methotrexate for at least 8 weeks prior to the Baseline Visit.
* At the Screening and Baseline Visits, the subject must have at least 6 swollen and 9 tender/painful joints using the 66/68 joint count scale.
* At the Screening Visit, the subject must have a C - reactive protein of at least 1.2 mg/dL or an erythrocyte sedimentation rate of at least 28 mm/hr.
* If taking a systemic corticosteroid, the maintenance dose of prednisone, or its equivalent, must be stable for at least 4 weeks prior to the Baseline Visit, may not exceed 10 mg/day and the subject should continue on that stable dose throughout the study.
* If taking a non-steroidal anti-inflammatory drug for the treatment of rheumatoid arthritis, the maintenance dose of the non-steroidal anti-inflammatory drug must be stable for at least 4 weeks prior to the Baseline Visit, and should continue on that stable dose throughout the trial.
* Had a forced expiratory volume in one second and a forced vital capacity greater than 80% of predicted at screening.

Exclusion Criteria:

* Had been diagnosed with any type of arthritis at age 16 or younger.
* Had achieved greater than or equal to 20% response improvement in rheumatoid arthritis signs and symptoms according to the American College of Rheumatology criteria during the placebo lead-in period.
* Had a history of a clinically significant illness, medical condition, or laboratory abnormality within 3 months prior to the Baseline Period that, in the investigator's opinion, would preclude the subject's participation in the study.
* Had a known history of human immunodeficiency virus infection.
* Had a known history of hepatitis B or C.
* Had uncontrolled hypertension.
* Had moderate or severe liver disease, as defined by one or more of the following at the Screening Visit:

  * Aspartate or alanine transaminase greater than 1.2 times the upper limit of normal.
  * Total bilirubin greater than 1.2 times the upper limit of normal (excluding subject's diagnosed with Gilbert's Disease).
  * Alkaline phosphatase greater than 1.5 times the upper limit of normal.
* Had elevated serum creatinine level for age and gender at the Screening Visit.
* Had hemoglobin less than 9.0 mg/dL, white blood cell count of less than 3000/mm3 or a platelet count less than 100,000/mm3 at the Screening Visit.
* Had an American College of Rheumatology revised rheumatoid arthritis functional status of IV at the Screening Visit.
* Was required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of TAK-783, including:

  * Disease-modifying antirheumatic drugs or biologic agents other than methotrexate in the 12 weeks prior to the Baseline Visit, including:

    * Sulfasalazine
    * Tetracycline
    * Leflunomide (AravaÒ)
    * Infliximab (RemicadeÒ)
    * Etanercept (EnbrelÒ)
    * Adalimumab (HumiraÒ)
    * Anakinra (KineretÒ)
  * Plaquenil in the 6 months prior to the Baseline Visit.
  * The subject has ever received abatacept (OrenciaÒ) or rituximab (RituxanÒ).
  * The subject has failed due to lack of efficacy with more than 2 disease-modifying antirheumatic drugs (other than methotrexate).
  * The subject has received any intra-articular, intramuscular, or intravenous corticosteroids within 4 weeks prior to the Baseline Visit.
  * The subject has had any previous use of cyclophosphamide, chlorambucil, or other alkylating agent.
  * Controlled-release oxycodone (OxyContinÒ) and other non-nonsteroidal anti-inflammatory drug long-acting analgesics.
  * Aspirin and aspirin-containing combination products used for analgesia. (Aspirin less than or equal to 325 mg/day for cardiac prophylaxis is permitted.)
* Was at high risk of an opportunistic infection because of a compromised immune system, in the investigator's opinion, with the exception of subjects receiving chronic steroid treatment.
* Had a history of, or a current inflammatory condition with signs and symptoms that might confound the diagnosis of rheumatoid arthritis (eg, connective tissue disease, systemic lupus erythematosis, psoriasis, psoriatic arthritis, spondyloarthropathy).
* Had been diagnosed as having a secondary, non-inflammatory type of arthritis (eg, osteoarthritis or fibromyalgia) that, in the investigator's opinion, is symptomatic enough to interfere with the evaluation of the efficacy of the study medications on the subject's primary diagnosis of rheumatoid arthritis.
* Had a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Had a body mass index greater than 35 at Screening.
* Had a previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug.
* Had received any investigational compound within 30 days prior to Randomization.
* Had donated more than 400 mL of blood within the 90 days preceding the beginning of the study.
* Had a known hypersensitivity to TAK 783 or its constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with greater than or equal to 20% improvement in Arthritis Signs and Symptoms according to the American College of Rheumatology | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Treatment-emergent adverse events. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Vital signs. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Electrocardiogram findings. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Spirometry tests. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Hematology Laboratory tests. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Chemistry Laboratory tests. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Urinalysis Laboratory tests. | Weeks 2, 4, 8, and 12 or Final Visit.

SECONDARY OUTCOMES:
Percent of subjects with greater than or equal to 50% improvement in Arthritis Signs and Symptoms according to the American College of Rheumatology | Weeks 2, 4, 8, and 12 or Final Visit.
Percent of subjects with greater than or equal to 70% improvement in Arthritis Signs and Symptoms according to the American College of Rheumatology | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in individual Arthritis Signs and Symptoms according to the American College of Rheumatology. | Weeks 2, 4, 8, and 12 or Final Visit.
Percent change from Baseline in the disability index of the Heath Assessment Questionnaire, based on the American College of Rheumatology criteria. | Weeks 2, 4, 8, and 12 or Final Visit.
Percent Change from Baseline in 36-Item Short-Form Quality of Life Assessments | Weeks 4 and 12 or Final Visit.
Change from Baseline in Swollen Joint Counts. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Tender Joint Counts. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Patient's Assessment of Pain. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Patient's Global Assessment of Disease Activity. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Physician's Global Assessment of Disease Activity. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Health Assessment Questionnaire. | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in Erythrocyte Sedimentation rate | Weeks 2, 4, 8, and 12 or Final Visit.
Change from Baseline in C-reactive Protein | Weeks 2, 4, 8, and 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (25):
- Czechia (6):
  - Brno-Bohunice
  - Hlučín
  - Pilsen
  - Prague
  - Uherské Hradiště
  - Zlín
- Latvia (2):
  - Daugavpils
  - Riga
- Romania (2):
  - Bucharest
  - Timișoara
- Russia (7):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Yaroslavl
  - Yekaterinburg
- Slovakia (6):
  - Košice
  - Martin
  - Nové Zámky
  - Piešťany
  - Poprad
  - Trnava
- Ukraine (2):
  - Donetsk
  - Kyiv